CLINICAL TRIAL: NCT01477528
Title: Study of Reduced Anti-coagulation/Anti-platelet Therapy in Patients With the HeartMate II LVAS (TRACE)
Brief Title: Study of Reduced Anti-coagulation/Anti-platelet Therapy in Patients With the HeartMate II Left Ventricular Assist System (LVAS) (TRACE)
Acronym: TRACE
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: TC-081611
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Anticoagulation; Left Ventricular Assist Device
Keywords: HeartMate II; Anticoagulation; Thoratec Corporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to obtain multi-center data on HeartMate II (HMII) patients managed with reduced anticoagulation or anti-platelet regimes, and the incidence of thrombotic and bleeding adverse events associated with these regimes.

ELIGIBILITY:
Inclusion Criteria:

* HeartMate II Left Ventricular Assist Device (LVAD) patient
* Patient has signed an informed consent for data collection.
* Patient was discharged, or is being discharged, from the hospital after their initial LVAD implant surgery.
* Patient:

  * at time of enrolling in study, is currently on, with the intention of being maintained on reduced anti-thrombotic therapy (RT) for chronic long-term management.

OR

-- On or after January 1, 2011 patient was being maintained on, or had been initiated with the intention of being maintained on, reduced anti-thrombotic therapy (RT) for chronic long-term management; but where RT was subsequently discontinued due to an adverse event or transplant, explant, or death.

Exclusion Criteria:

* Patients under acute management of anti-thrombotic agents before a final decision on long term antithrombotic strategy.
* Patients requiring a legal representative to sign consent form, rather than themselves.
* Patient is being managed on other anti-thrombotic agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HeartMate II VAD that are on reduced anticoagulation/antiplatelet regimine
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Rate of thromboembolic events and hemorrhagic events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec Europe Limited; David Farrar, PhD, Study Director — Thoratec Corporation
Locations (18):
- United States (9):
  - Sharp Memorial Hospital, San Diego, California
  - University of Florida (Shands), Gainesville, Florida
  - Advocate Christ Hospital, Oak Lawn, Illinois
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
- Medical University of Vienna, Vienna, Austria
- IKEM, Prague, Czechia
- France (5):
  - Service de Chirurgie Cardiaque, Grenoble
  - Hopital Cardiologique, Lille
  - Chirurgie Thoracique et Cardiovasculaire Groupe hospitalier Pitie-Salpetriere, Paris
  - Hôpital Pontchaillou, Rennes
  - Charles Nicolle University Hospital, Rouen
- Germany (2):
  - University of Freiburg Medical Center, Freiburg im Breisgau
  - Medical University Hannover, Hanover